CLINICAL TRIAL: NCT01716988
Title: Pharmacokinetics of Micafungin in Critically Ill Patients With Invasive Candidiasis
Brief Title: Pharmacokinetics of Micafungin in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Jan-Willem C Alffenaar, PharmD, PhD, University Medical Center Groningen
Other Study IDs: NL39246.042.12
Record Dates: First submitted 2012-10-08; First posted 2012-10-30 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Critical Illness; Invasive Candidiasis
Keywords: Micafungin; pharmacokinetics; invasive candidiasis; intensive care
MeSH Terms: conditions — Critical Illness; Candidiasis, Invasive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Micafungin

SUMMARY:
A study of micafungin in ICU versus non-ICU patients showed a significantly lower treatment success in ICU patients compared with non-ICU patients. It is known that in critically ill patients, alterations in function of various organs and body systems can influence the pharmacokinetics and hence the plasma concentration of a drug. The pharmacokinetic parameters of micafungin in critically ill patients are most likely different, but this has not been specifically studied.

The pharmacokinetic parameters of micafungin in critically ill patients will be established and plasma concentrations of micafungin will be correlated with disease severity.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with micafungin.
* Admission to an ICU.
* Age ≥ 18 years.
* Invasive candidiasis.

Exclusion Criteria:

* Blood sampling not possible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with invasive candidiasis admitted to an intensive care unit.
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2012-10; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Correlation of pharmacokinetic parameters/plasma concentrations of micafungin with disease severity. | 4 days
  Correlation of the level of micafungin concentration with disease severity scores. Correlation of pharmacokinetic parameters (clearance, half-life) of micafungin with disease severity scores.

SECONDARY OUTCOMES:
Pharmacokinetic parameters of micafungin in ICU patients. | 4 days
  Calculate the pharmacokinetic parameters (clearance, half life, volume of distribution) of micafungin.
Time (in days) to culture conversion. | max 28 days
  Number of days untill cultures are negative.
Correlation of the plasma concentration of micafungin with response to treatment. | max 28 days
  Correlation of the level of micafungin concentration with outcome.
Correlation of the plasma concentration of micafungin with inflammation parameters. | 4 days
  Correlation of the level of micafungin concentration with interleukin-6, interleukin-8 and procalcitonin.
Area under the concentration-time curve (AUC)/minimal inhibitory concentration (MIC) ratio. | max 28 days
  Area under the concentration-time curve of micafungin devided by the minimal inhibitory concentration of the candida species.
Composing a pharmacokinetic model of micafungin in critically ill patients. | max 28 days
  Composing a pharmacokinetic model of micafungin to estimate the 24-hours AUC of micafungin based on limited samples.
Highest observed plasma concentration (Cmax)/minimal inhibitory concentration (MIC) ratio. | 28 days
  Highest observed plasma concentration of micafungin devided by the minimal inhibitory concentration of the candida species.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Boonstra JM, van der Elst KC, Veringa A, Jongedijk EM, Bruggemann RJ, Koster RA, Kampinga GA, Kosterink JG, van der Werf TS, Zijlstra JG, Touw DJ, Alffenaar JWC. Pharmacokinetic Properties of Micafungin in Critically Ill Patients Diagnosed with Invasive Candidiasis. Antimicrob Agents Chemother. 2017 Nov 22;61(12):e01398-17. doi: 10.1128/AAC.01398-17. Print 2017 Dec. PMID 28971861